CLINICAL TRIAL: NCT04224090
Title: Diagnostic Performance of a Rational and Standardized New Method for the Echocardiographic
Brief Title: Diagnostic Performance of a New Method for the Echocardiographic Assessment of Coronary Arteries Abnormalities
Status: Completed | Type: Observational
Sponsor: ITAB - Institute for Advanced Biomedical Technologies (Other)
Collaborators: Ospedali Riuniti Ancona (Other)
Responsible Party: Principal Investigator, Francesco Bianco, Researcher, ITAB - Institute for Advanced Biomedical Technologies
Other Study IDs: Cor001
Record Dates: First submitted 2020-01-08; First posted 2020-01-13 (Actual); Last update posted 2022-01-24 (Actual); Status verified 2022-01

CONDITIONS: Coronary Artery Anomaly
Keywords: Coronary arteries abnormalities; Coronary arteries anomaly; Coronary origin from the wrong sinus of Valsalva; Echocardiography

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Congenita coronary abnormalities (CAA): All the coronary arteries were differing from the definition of "normal": when do not arise from the appropriate sinus of Valsalva (right or left) and not present a proper course and termination.
  Interventions: Diagnostic Test: Echocardiographic assessment of coronary arteries origin and proximal course

INTERVENTIONS:
Diagnostic Test: Echocardiographic assessment of coronary arteries origin and proximal course — Echocardiographic assessment of CAA utilizing 4 specific echocardiographic acoustic windows: parasternal short-axis (PSAX), parasternal long-axis (PLAX), apical 4/5-chambers views.

SUMMARY:
Coronary artery anomalies (CAA) are a rare congenital condition, accounting abnormalities of origin, course, destination, size, and number of the coronary vessels. In normal hearts, the coronary arteries, the left and right coronary arteries (LCA and RCA, respectively) originate from the two facing aortic sinuses of Valsalva, so-called left and right. To overcome the echocardiographic limitations, the investigators designed, studied and implemented in our Institute a specific echocardiographic-based two-dimensional non-Doppler 4-views approach for the diagnosis of CAA.

DETAILED DESCRIPTION:
The method consisted of 4-CAA-focused specific views, routinely available from any echocardiographic exam: parasternal short-axis (PSAX), parasternal long-axis (PLAX), apical 4/5-chambers views. PSAX, the traditional approach, along with the PLAX, and the apical 4/5-chambers views.

A hallmark of CAA was considered the absence of a proper visualization of the origin of the coronary arteries from the aortic root. In addition, the presence of the ring sign, visualized from the PLAX was considered as abnormal. This sign is of interest when an aberrant left or right CAA is suspected. A coronary artery originating from the contralateral aortic sinus, along its intramural course, crosses the mid-anterior line of the circular aorta to reach the sinus of Valsalva of its intended origin. Consequently, its cross-section should be visible in an orthogonal view traversing the mid-long axis of the aorta, namely the parasternal long-axis view.

ELIGIBILITY:
Inclusion Criteria:

* patients undergoing their first echocardiographic examination

Exclusion Criteria:

* already known congenital heart disease and cardiomyopathies

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Outpatients (neonates, pediatrics, adolescents and young adults) undergoing routine echocardiography in our department
Sampling Method: Non-Probability Sample
Enrollment: 4000 (Actual)
Dates: Start 2014-01-01 (Actual); Primary Completion 2020-12-01 (Actual); Study Completion 2021-12-01 (Actual)

PRIMARY OUTCOMES:
CAA | At the time of the routine echocardiography assessment
  The number of coronary arteries anomalies echocardiographically detected

CONTACTS AND LOCATIONS:
Overall Officials: Francesco Bianco, M.D., Principal Investigator — Ospedali Riuniti
Locations (1):
- Ospedali Riuniti, Ancona, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Cheezum MK, Liberthson RR, Shah NR, Villines TC, O'Gara PT, Landzberg MJ, Blankstein R. Anomalous Aortic Origin of a Coronary Artery From the Inappropriate Sinus of Valsalva. J Am Coll Cardiol. 2017 Mar 28;69(12):1592-1608. doi: 10.1016/j.jacc.2017.01.031. PMID 28335843
- [Background] Angelini P. Normal and anomalous coronary arteries in humans. In. Coronary artery anomalies: A comprehensive approach. Philadelphia: Lippincott Williams & Wilkins; 1999.
- [Background] Perez-Pomares JM, de la Pompa JL, Franco D, Henderson D, Ho SY, Houyel L, Kelly RG, Sedmera D, Sheppard M, Sperling S, Thiene G, van den Hoff M, Basso C. Congenital coronary artery anomalies: a bridge from embryology to anatomy and pathophysiology--a position statement of the development, anatomy, and pathology ESC Working Group. Cardiovasc Res. 2016 Feb 1;109(2):204-16. doi: 10.1093/cvr/cvv251. Epub 2016 Jan 11. PMID 26811390
- [Background] Basso C, Maron BJ, Corrado D, Thiene G. Clinical profile of congenital coronary artery anomalies with origin from the wrong aortic sinus leading to sudden death in young competitive athletes. J Am Coll Cardiol. 2000 May;35(6):1493-501. doi: 10.1016/s0735-1097(00)00566-0. PMID 10807452
- [Background] Maron BJ, Doerer JJ, Haas TS, Tierney DM, Mueller FO. Sudden deaths in young competitive athletes: analysis of 1866 deaths in the United States, 1980-2006. Circulation. 2009 Mar 3;119(8):1085-92. doi: 10.1161/CIRCULATIONAHA.108.804617. Epub 2009 Feb 16. PMID 19221222
- [Background] Lang RM, Badano LP, Mor-Avi V, Afilalo J, Armstrong A, Ernande L, Flachskampf FA, Foster E, Goldstein SA, Kuznetsova T, Lancellotti P, Muraru D, Picard MH, Rietzschel ER, Rudski L, Spencer KT, Tsang W, Voigt JU. Recommendations for cardiac chamber quantification by echocardiography in adults: an update from the American Society of Echocardiography and the European Association of Cardiovascular Imaging. J Am Soc Echocardiogr. 2015 Jan;28(1):1-39.e14. doi: 10.1016/j.echo.2014.10.003. PMID 25559473
- [Background] Jureidini SB, Marino CJ, Singh GK, Balfour IC, Rao PS, Chen SC. Aberrant coronary arteries: a reliable echocardiographic screening method. J Am Soc Echocardiogr. 2003 Jul;16(7):756-63. doi: 10.1016/S0894-7317(03)00321-3. PMID 12835663
- [Background] Brown LM, Duffy CE, Mitchell C, Young L. A practical guide to pediatric coronary artery imaging with echocardiography. J Am Soc Echocardiogr. 2015 Apr;28(4):379-91. doi: 10.1016/j.echo.2015.01.008. Epub 2015 Feb 15. PMID 25691000
- [Derived] Bianco F, Colaneri M, Bucciarelli V, Surace FC, Iezzi FV, Primavera M, Biasi A, Giusti G, Berton E, Baldoni M, Renda G, Baldinelli A, Gallina S, Pozzi M. Echocardiographic screening for the anomalous aortic origin of coronary arteries. Open Heart. 2021 Jan;8(1):e001495. doi: 10.1136/openhrt-2020-001495. PMID 33431619